CLINICAL TRIAL: NCT01603056
Title: A Randomised, Double-blind, Placebo-controlled Phase III Multicentre Clinical Trial Investigating the Efficacy and Safety of Pangramin SLIT HDM-mix in Chinese Population With House Dust Mite Induced Rhinitis With or Without Asthma.
Brief Title: Efficacy and Safety Trial of Pangramin SLIT HDM-mix in Subjects With House Dust Mite Induced Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PS-M-01
Record Dates: First submitted 2012-04-27; First posted 2012-05-22 (Estimated); Results first posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-03

CONDITIONS: Allergic Rhinitis
Keywords: House dust mite induced allergic rhinitis.
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PANGRAMIN SLIT HDM MIX (Experimental): PANGRAMIN SLIT HDM MIX Up-dosing phase (vial 0 to vial 4) + maintenance phase (3 times per week), for 12 months.
  Interventions: Biological: Pangramin SLIT HDM mix.
- Placebo (Placebo Comparator): Placebo Up-dosing phase (vial 0 to vial 4) + maintenance phase (3 times per week), for 12 months.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Pangramin SLIT HDM mix. — Up-dosing phase (vial 0 to vial 4) + maintenance phase (3 times per week), for 12 months.
  Arms: PANGRAMIN SLIT HDM MIX
Biological: Placebo — Up-dosing phase (vial 0 to vial 4) + maintenance phase (3 times per week), for 12 months.
  Arms: Placebo

SUMMARY:
Primary aim is to evaluate the efficacy of specific immunotherapy with Pangramin SLIT HDM-mix compared to placebo in the treatment of House Dust Mite (HDM) induced rhinitis with or without asthma.

Sublingual immunotherapy has been used during several years and has been shown to provide benefits compare to traditional subcutaneous treatment. This study will investigate if improvements in rhinitis symptoms and less use of symptomatic medication can be obtained as a consequence of being treated under specific immunotherapy.

This study aim also to contribute to the documentation of tolerability and safety profile of Pangramin HDM Mix.

DETAILED DESCRIPTION:
Extensive clinical experience has been gained due to the widespread use of Pangramin® SLIT and other SLIT products as named patient products, both with respect to the types and the frequencies of the adverse events(AEs) observed. No safety concerns have been found.

The optimal therapeutic dose range regarding SLIT is not fully elucidated. The fate of the allergen after sublingual administration is not known in detail, i.e. to what extent is the allergen absorbed over the mucosa or swallowed and how this is related to volume, excipients etc. The relationship between dose and effect is thus not fully elucidated. The general recommendation is to use a dose inducing a clinical relevant effect in most patients without causing unacceptable adverse events. As Pangramin SLIT HDM-mix has a safety profile that allows a single daily intake by the patient at home, the dosage at this trial will be the same as marketed product.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 5 to ≤ 55 years of age.
* A history HDM induced allergic rhinitis.
* Use of medication for the control of rhinoconjunctivitis symptoms.
* Positive Skin Prick Test (SPT).
* Positive specific IgE.

Exclusion Criteria:

* PEF ≤ 70% of predicted value.
* History of significant symptomatic seasonal or perennial allergic rhinitis and/or asthma caused by an allergen to which the patient is regularly exposed, and sensitized (e.g. pollens, cat, dog, cockroach…except house dust mites).
* Severe asthma.
* Current symptoms of upper respiratory tract infection or other relevant infectious process.
* Current food allergies with oral allergy syndrome.
* A clinical history of chronic sinusitis.
* Current severe atopic dermatitis.
* Concomitant or previous treatment by immunotherapy.

Ages: 5 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 617 (Actual)
Dates: Start 2009-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Luo, Professor, Principal Investigator — Beijing Tongren Hospital
Locations (1):
- No.2, Chongwenmennei Street, Dongcheng District, Beijing, Beijing Municipality, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PANGRAMIN SLIT HDM MIX | Placebo
Started | 413 | 204
Completed | 379 | 190
Not Completed | 34 | 14

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | PANGRAMIN SLIT HDM MIX | Placebo | Total
Number analyzed (Participants) | 400 | 200 | 600
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.74 (12.98) | 19.47 (12.01) | 20.31 (12.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 87 | 259
  Male | 228 | 113 | 341
Region of Enrollment [Number; unit: participants]
  China | 400 | 200 | 600

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline in Rhinoconjunctivitis Symptoms Score at 11 - 12 Months Between the Actively Treated Patients and the Placebo Treated.
Description: Subjects completed symptom assessments and recorded the results in the patient diary cards on a daily basis. A total of six rhinoconjunctivitis symptoms were measured on a scale from 0-3 as follows:
  0 = No symptoms.
  1. = Mild symptoms.
  2. = Moderate symptoms. 3= Severe symptoms.
  The six symptoms are classified in 2 groups as follows:
  Nose symptoms: Runny nose, Blocked nose, Sneezing, Itchy nose; Eye symptoms: Gritty feeling/red/itchy eyes, Watery eyes. The six symptom scores were summed to obtain the rhinoconjunctivitis symptoms score with range 0(best) to 18(worst).
  Baseline was set as 8 weeks before randomization as from V1 (Week -8) to V2 (Week 0). 11-12months' end evaluation period was set from V8(Week 44) to V9(Week 52). These two average rhinoconjunctivitis symptoms scores (Baseline and 11-12months) were calculated for each patient as the sum of the daily score throughout the 2 months(8 weeks in count) in evaluation period and divided with the days with diary.
Time Frame: Baseline: From V1 date(Week -8) to V2 date(Week 0); 11-12months: From V8 date(Week 44) to V9 date(Week 52).
Population: The analysis was performed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale (Symptom Score)
Arm/Group | PANGRAMIN SLIT HDM MIX | Placebo
Number analyzed (Participants) | 400 | 200
units on a scale (Symptom Score) | -1.77 (2.13) | -1.83 (2.18)
Statistical Analysis 1: Comparison: PANGRAMIN SLIT HDM MIX vs Placebo; Test type: Superiority or Other; p = 0.743, t-test, 2 sided

2. Primary Outcome: The Change From Baseline in Rhinoconjunctivitis Medication Score at 11 - 12 Months Between the Actively Treated Patients and the Placebo Treated.
Description: Subjects were provided with open-labelled rescue medication to be used as needed for treatment of their rhinoconjunctivitis symptoms. Subjects reported their use of specific rescue medication via the patient diary cards. Scoring principles were applied to transform the number of rescue medication doses used into medication scores.The scores of all the medication used were summed to produce the daily rhinoconjunctivitis medication score range from 0 to 32. A lower medication score means the patient use less medication, and represent a better outcome; on the contrary, a higher medication score means the patient use more medication, and represent a worse outcome.
  Baseline was from V1 (Week -8) to V2 (Week 0). The end evaluation period was set from V8(Week 44) to V9(Week 52). These two average scores (Baseline and End) were calculated for each patient as the sum of the daily score throughout the 2 months(8 weeks in count) in evaluation period and divided with the days in diary.
Time Frame: Baseline: From V1 date(Week -8) to V2 date(Week 0); 11-12months: From V8 date(Week 44) to V9 date(Week 52).
Population: The analysis was performed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale (Medication Score)
Arm/Group | PANGRAMIN SLIT HDM MIX | Placebo
Number analyzed (Participants) | 400 | 200
units on a scale (Medication Score) | -2.17 (2.77) | -2.16 (2.77)
Statistical Analysis 1: Comparison: PANGRAMIN SLIT HDM MIX vs Placebo; Test type: Superiority or Other; p = 0.627, t-test, 2 sided

3. Secondary Outcome: The Change From Baseline in Rhinitis Symptom Score at 11 - 12 Months Between the Actively Treated Patients and the Placebo Treated.
Description: Subjects were instructed by the investigator on how to complete symptom assessments and recorded the results in the patient diary cards on a daily basis.
  A total of 4 rhinitis symptoms were measured on a scale from 0-3 as follows:
  0 = No symptoms.
  1. = Mild symptoms.
  2. = Moderate symptoms. 3= Severe symptoms. The 4 symptoms are as follows: Runny nose, Blocked nose, Sneezing, Itchy nose. The 4 symptom scores were summed to obtain the rhinitis symptoms score with range 0(best) to 12(worst).
  Baseline was set as 8 weeks before randomization as from V1 (Week -8) to V2 (Week 0). 11-12months' end evaluation period was set from V8(Week 44) to V9(Week 52). These two average scores (Baseline and 11-12months) were calculated for each patient as the sum of the daily score throughout the 2 months(8 weeks in count) in evaluation period and divided with the days with diary.
Time Frame: Baseline: From V1 date(Week -8) to V2 date(Week 0); 11-12months: From V8 date(Week 44) to V9 date(Week 52).
Population: The analysis was performed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale (Symptom score)
Arm/Group | PANGRAMIN SLIT HDM MIX | Placebo
Number analyzed (Participants) | 400 | 200
units on a scale (Symptom score) | -1.44 (1.78) | -1.48 (1.78)
Statistical Analysis 1: Comparison: PANGRAMIN SLIT HDM MIX vs Placebo; Test type: Superiority or Other; p = 0.74, t-test, 2 sided

4. Secondary Outcome: The Change From Baseline in Conjunctivitis Symptom Score at 11 - 12 Months Between the Actively Treated Patients and the Placebo Treated.
Description: Subjects were instructed by the investigator on how to complete symptom assessments and recorded the results in the patient diary cards on a daily basis.
  A total of 2 conjunctivitis symptoms were measured on a scale from 0-3 as follows:
  0 = No symptoms.
  1. = Mild symptoms.
  2. = Moderate symptoms. 3= Severe symptoms. The 2 symptoms as follows: Gritty feeling/red/itchy eyes, Watery eyes. The 2 symptom scores were summed to obtain the conjunctivitis symptoms score with range 0(best) to 6(worst).
  Baseline was set as 8 weeks before randomization as from V1 (Week -8) to V2 (Week 0). 11-12months' end evaluation period was set from V8(Week 44) to V9(Week 52). These two average scores (Baseline and 11-12months) were calculated for each patient as the sum of the daily score throughout the 2 months(8 weeks in count) in evaluation period and divided with the days with diary.
Time Frame: Baseline: From V1 date(Week -8) to V2 date(Week 0); 11-12months: From V8 date(Week 44) to V9 date(Week 52).
Population: The analysis was performed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale(Symptom score)
Arm/Group | PANGRAMIN SLIT HDM MIX | Placebo
Number analyzed (Participants) | 400 | 200
units on a scale(Symptom score) | -0.36 (0.61) | -0.38 (0.71)
Statistical Analysis 1: Comparison: PANGRAMIN SLIT HDM MIX vs Placebo; Test type: Superiority or Other; p = 0.641, t-test, 2 sided

5. Secondary Outcome: The Change From Baseline in Asthma Symptom Score at 11 - 12 Months Between the Actively Treated Patients and the Placebo Treated.
Description: Subjects were instructed by the investigator on how to complete symptom assessments and recorded the results in the patient diary cards on a daily basis.
  A total of 4 Asthma symptoms were measured on a scale from 0-3 as follows:
  0 = No symptoms.
  1. = Mild symptoms.
  2. = Moderate symptoms. 3= Severe symptoms. The 4 symptoms as follows: Cough, Wheeze, Chest tightness/shortness of breath (dyspnoea), Exercise induced symptoms. The 4 symptom scores were summed to obtain the asthma symptoms score with range 0(best) to 12(worst).
  Baseline was set as 8 weeks before randomization as from V1 (Week -8) to V2 (Week 0). 11-12months' end evaluation period was set from V8(Week 44) to V9(Week 52). These two average scores (Baseline and 11-12months) were calculated for each patient as the sum of the daily score throughout the 2 months(8 weeks in count) in evaluation period and divided with the days with diary.
Time Frame: Baseline: From V1 date(Week -8) to V2 date(Week 0); 11-12months: From V8 date(Week 44) to V9 date(Week 52).
Population: The analysis was performed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale(Symptom score)
Arm/Group | PANGRAMIN SLIT HDM MIX | Placebo
Number analyzed (Participants) | 400 | 200
units on a scale(Symptom score) | -0.36 (0.82) | -0.35 (0.75)
Statistical Analysis 1: Comparison: PANGRAMIN SLIT HDM MIX vs Placebo; Test type: Superiority or Other; p = 0.818, t-test, 2 sided

6. Secondary Outcome: Percentage of Healthy Days in This Study Between the Actively Treated Patients and the Placebo Treated.
Description: A healthy day is a day without rhinoconjunctivitis symptoms and without any intake of rescue medication. Percentage of healthy days is the healthy days of subject in this study divided by the total study days.
Time Frame: Total study year
Population: The analysis was performed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: Percentage of healthy days
Arm/Group | PANGRAMIN SLIT HDM MIX | Placebo
Number analyzed (Participants) | 400 | 200
Percentage of healthy days | 21.92 (31.8) | 18.85 (30.33)
Statistical Analysis 1: Comparison: PANGRAMIN SLIT HDM MIX vs Placebo; Test type: Superiority or Other; p = 0.391, t-test, 2 sided

7. Secondary Outcome: The Change From Baseline in Nasal Complain Scores on Visual Analog Scale at 11-12 Months Between the Actively Treated Patients and the Placebo Treated.
Description: The average rhinoconjunctivitis VAS score (baseline to first year). The scale answers the question 'How have your nasal complaints been today?' from 0 = no symptoms to 10 = severe symptoms.
  The baseline VAS rhinoconjunctivitis score is the average value of VAS scores in V1 (Screen Visit, Week -8) and V2 (Randomization visit, Week 0), and Evaluation period (Months 11-12) VAS rhinoconjunctivitis score is the average value of VAS scores in V8 (Week 44) and V9 (Week 52).
Time Frame: Baseline: From V1 date(Week -8) to V2 date(Week 0); 11-12months: From V8 date(Week 44) to V9 date(Week 52).
Population: The analysis was performed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale (VAS Score)
Arm/Group | PANGRAMIN SLIT HDM MIX | Placebo
Number analyzed (Participants) | 400 | 200
units on a scale (VAS Score) | -2.45 (1.92) | -2.33 (2.13)
Statistical Analysis 1: Comparison: PANGRAMIN SLIT HDM MIX vs Placebo; Test type: Superiority or Other; p = 0.497, t-test, 2 sided

8. Secondary Outcome: The Change From Baseline in Rhinitis Quality of Life Questionnaire at 12 Months Between the Actively Treated Patients and the Placebo Treated.
Description: The baseline RQLQ value was collected in Visit 1 (Week -8) and the 12 months' RQLQ value was collected in Visit 9 (Week 52).
  The maximum value of RQLQ score is 168 and the minimum one is 0. The score is decreased as the life quality is better.
Time Frame: Visit 1 date(Week -8), Visit 9 date(Week 52).
Population: The analysis was performed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale (RQLQ score)
Arm/Group | PANGRAMIN SLIT HDM MIX | Placebo
Number analyzed (Participants) | 400 | 200
units on a scale (RQLQ score) | -0.87 (1.07) | -0.75 (1.01)
Statistical Analysis 1: Comparison: PANGRAMIN SLIT HDM MIX vs Placebo; Test type: Superiority or Other; p = 0.222, t-test, 2 sided

9. Secondary Outcome: Global Assessment of Rhinoconjunctivitis Symptom After Treatment Between the Actively Treated Patients and the Placebo Treated.
Description: Comparing overall rhinoconjunctivitis symptoms at the end of study year Between the Actively Treated Patients and the Placebo Treated.
Time Frame: Visit 9 date, Week 52
Population: The analysis was performed in the Full Analysis Set.
Measure: Number; unit: participants
Arm/Group | PANGRAMIN SLIT HDM MIX | Placebo
Number analyzed (Participants) | 400 | 200
participants
  Great | 72 | 39
  Good | 213 | 91
  Fair | 93 | 58
  Worse | 5 | 3
  Not Done | 17 | 9
Statistical Analysis 1: Comparison: PANGRAMIN SLIT HDM MIX vs Placebo; Test type: Superiority or Other; p = 0.438, Fisher Exact

10. Secondary Outcome: The Change From Baseline in Rhinitis Medication Score at 11 - 12 Months Between the Actively Treated Patients and the Placebo Treated.
Description: Subjects were provided with open-labelled rescue medication to be used as needed for treatment of their Rhinitis symptoms. Subjects reported their use of specific rescue medication via the patient diary cards. Scoring principles were applied to transform the number of rescue medication doses used into medication scores. The scores of all the medication used were summed to produce the daily Rhinitis medication score range from 0 to 30. A lower medication score means the patient use less medication, and represent a better outcome; on the contrary, a higher medication score means the patient use more medication, and represent a worse outcome.
  Baseline was set as from V1 (Week -8) to V2 (Week 0). 11-12months' end evaluation period was set from V8(Week 44) to V9(Week 52). These two average scores (Baseline and 11-12months) were calculated for each patient as the sum of the daily score throughout the 2 months(8 weeks in count) in evaluation period and divided with the days with diary.
Time Frame: Baseline: From V1 date(Week -8) to V2 date(Week 0); 11-12months: From V8 date(Week 44) to V9 date(Week 52).
Population: The analysis was performed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale(Medication score)
Arm/Group | PANGRAMIN SLIT HDM MIX | Placebo
Number analyzed (Participants) | 400 | 200
units on a scale(Medication score) | -2.16 (2.7) | -2.19 (2.7)
Statistical Analysis 1: Comparison: PANGRAMIN SLIT HDM MIX vs Placebo; Test type: Superiority or Other; p = 0.465, t-test, 2 sided

11. Secondary Outcome: The Change From Baseline in Asthma Quality of Life Questionnaire at 12 Months Between the Actively Treated Patients and the Placebo Treated.
Description: The baseline AQLQ value was collected in Visit 1 (Week -8) and the 12 months' RQLQ value was collected in Visit 9 (Week 52). The maximum value of RQLQ score is 217 and the minimum one is 0. The score is elevated as the life quality is better.
Time Frame: Visit 1 date(Week -8), Visit 9 date(Week 52).
Population: The analysis was performed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale(AQLQ score)
Arm/Group | PANGRAMIN SLIT HDM MIX | Placebo
Number analyzed (Participants) | 400 | 200
units on a scale(AQLQ score) | 0.33 (0.9) | 0.25 (1.04)
Statistical Analysis 1: Comparison: PANGRAMIN SLIT HDM MIX vs Placebo; Test type: Superiority or Other; p = 0.123, t-test, 2 sided

12. Secondary Outcome: The Change From Baseline in Asthma Medication Score at 11 - 12 Months Between the Actively Treated Patients and the Placebo Treated
Description: Subjects were provided with open-labelled rescue medication to be used as needed for treatment of their Asthma symptoms. Subjects reported their use of specific rescue medication via the patient diary cards. Scoring principles were applied to transform the number of rescue medication doses used into medication scores. The scores of all the medication used were summed to produce the daily asthma medication score range from 0 to 32. A lower medication score means the patient use less medication, and represent a better outcome; on the contrary, a higher medication score means the patient use more medication, and represent a worse outcome.
  Baseline was set as from V1 (Week -8) to V2 (Week 0). 11-12months' end evaluation period was set from V8(Week 44) to V9(Week 52). These two average scores (Baseline and 11-12months) were calculated for each patient as the sum of the daily score throughout the 2 months in evaluation period and divided with the days with diary.
Time Frame: Baseline: From V1 date(Week -8) to V2 date(Week 0); 11-12months: From V8 date(Week 44) to V9 date(Week 52).
Population: The analysis was performed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale(Medication score)
Arm/Group | PANGRAMIN SLIT HDM MIX | Placebo
Number analyzed (Participants) | 400 | 200
units on a scale(Medication score) | -0.15 (1.34) | -0.09 (0.97)
Statistical Analysis 1: Comparison: PANGRAMIN SLIT HDM MIX vs Placebo; Test type: Superiority or Other; p = 0.719, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: All events meeting the definition of an adverse event must be collected and reported from the first trial-related activity after the patient signs the informed consent and until follow up telephone contact. The reporting time frame is almost one year.
Description: The analysis was performed in the Safety Set.
Arm/Group | PANGRAMIN SLIT HDM MIX | Placebo
Serious Adverse Events (participants affected / at risk) | 7/402 | 3/200
Other Adverse Events (participants affected / at risk) | 299/402 | 140/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PANGRAMIN SLIT HDM MIX (N=402) | Placebo (N=200)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Acute bronchial asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Left ureteral calculi (Surgical and medical procedures) | 1 (1) | 0 (0)
Acute purulent tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Deflection of nasal septum (Surgical and medical procedures) | 1 (1) | 0 (0)
Chronic hypertrophic rhinitis (Surgical and medical procedures) | 1 (1) | 0 (0)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PANGRAMIN SLIT HDM MIX (N=402) | Placebo (N=200)
Rhinopharyngitis (Infections and infestations) | 119 (207) | 52 (107)
Upper respiratory tract infection (Infections and infestations) | 90 (188) | 38 (86)
Asthma (Respiratory, thoracic and mediastinal disorders) | 48 (64) | 21 (39)
Cough (Respiratory, thoracic and mediastinal disorders) | 46 (84) | 20 (35)
Bronchitis (Infections and infestations) | 33 (54) | 21 (30)
Fever (General disorders) | 24 (34) | 18 (22)
Eye pruritus (Eye disorders) | 20 (24) | 11 (13)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 (61) | 6 (19)
Diarrhea (Gastrointestinal disorders) | 16 (25) | 9 (10)
Oropharyngeal (Respiratory, thoracic and mediastinal disorders) | 15 (21) | 6 (8)
Headache (Nervous system disorders) | 14 (16) | 2 (2)
Tonsillitis (Infections and infestations) | 11 (15) | 7 (10)
Erythra (Skin and subcutaneous tissue disorders) | 10 (11) | 4 (7)
Oral hypoesthesia (General disorders) | 9 (14) | 7 (7)
Chest discomfort (General disorders) | 9 (14) | 2 (2)
Conjunctivitis (Eye disorders) | 5 (6) | 7 (7)
Dental ulcer (Gastrointestinal disorders) | 8 (10) | 6 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (12) | 5 (6)
Odontalgia (Gastrointestinal disorders) | 5 (6) | 5 (6)
Gastritis (Gastrointestinal disorders) | 3 (3) | 6 (8)
Epigastric pain (Gastrointestinal disorders) | 5 (6) | 4 (10)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right to review and comment any manuscript within 30 days of receipt, but cannot prevent publications of findings. Sponsor will review the communications for accuracy (thus avoiding potential discrepancies with submissions to health authorities), verify that the confidential information is not being inadvertently divulged and provide any relevant supplementary information.